CLINICAL TRIAL: NCT02410551
Title: Pacritinib Prior to Transplant for Patients With Myeloproliferative Neoplasms (MPN)
Brief Title: Pacritinib Before Transplant for Myeloproliferative Neoplasms (MPN)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0786; NCI-2015-01123 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Myeloproliferative Diseases
Keywords: Myeloproliferative Diseases; Myeloproliferative Neoplasms; MPN; Myelofibrosis; Polycythemia vera; PV; Essential thrombocythemia; Allogeneic stem cell transplantation; Allo TP; Pacritinib; Busulfan; Busulfex; Myleran; Questionnaires; Surveys; Phone calls
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Polycythemia Vera; Thrombocythemia, Essential | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Busulfan; Surveys and Questionnaires; Stem Cell Transplantation; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pacritinib + Allogeneic Stem Cell Transplantation (Experimental): Participants start Pacritinib 200 mg by mouth twice a day. Participants proceed to transplant after 60 days of Pacritinib but not more than 180 days. Pacritinib stopped 21 days prior to starting preparative regimen for standard of care stem cell transplantation (SOC Allo TP). SOC transplant conditioning with Fludarabine and Busulfan AUC of 4000 microMol-min per day providing that pharmacokinetic can be done, otherwise Busulfan dose given as a fixed dose of 100 mg/m2 daily for four days. Questionnaires about symptoms and quality of life completed at baseline, 1, 3, 6, and 12 months after transplant. Phone calls made by study staff to participant on second and third week of each month.
  Interventions: Drug: Pacritinib; Drug: Busulfan; Behavioral: Questionnaires; Behavioral: Phone Calls; Procedure: Allogeneic Stem Cell Transplantation; Drug: Fludarabine

INTERVENTIONS:
Drug: Pacritinib — 200 mg by mouth twice a day for 60 days.
Drug: Busulfan — Busulfan AUC of 4000 microMol-min per day providing that pharmacokinetic can be done, otherwise Busulfan dose given as a fixed dose of 100 mg/m2 daily for four days.
  Other Names: Busulfex; Myleran
Behavioral: Questionnaires — Questionnaires completed at baseline, 1, 3, 6, and 12 months after transplant.
  Other Names: Surveys
Behavioral: Phone Calls — Phone calls made by study staff to participant on second and third week of each month.
Procedure: Allogeneic Stem Cell Transplantation — Allogeneic stem cell transplantation (Allo TP) 60 days after starting Pacritinib but not more than 180 days.
  Other Names: Stem cell transplant
Drug: Fludarabine — Fludarabine taken along with Busulfan as per standard of care as preparative regimen for allogeneic stem cell transplantation (Allo TP).
  Other Names: Fludarabine phosphate; Fludara

SUMMARY:
The goal of this clinical research study is to learn if giving pacritinib before standard of care drugs followed by an allogeneic stem cell transplant can help to control myeloproliferative neoplasms. The safety of this therapy will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will take pacritinib at about the same time each day by mouth, 2 times each day. Your doctor will tell you when to start and stop taking pacritinib. You may be able to take the drug for about 2-6 months depending on how you tolerate the drug and when your transplant date is. If you do not receive your transplant, you may be able to continue taking the study drug as long as the doctor thinks it is in your best interest.

You must swallow the capsules whole with a glass (about 8 ounces) of water. Do not open, break, or chew the capsules.

If you vomit or miss a dose of pacritinib, take your next dose of pacritinib at your regular time. Do not "make up" a missed or vomited dose.

You will be given a study drug diary to write down what time you take each dose of pacritinib. You need to bring the study drug diary, any leftover study drug, and any empty study drug containers with you to each study visit.

The dose of pacritinib you receive may be lowered or stopped, if the doctor thinks it is needed.

About 21 days after your last dose of pacritinib, you will given standard of care drugs and you will have an allogeneic stem cell transplant. Your doctor will explain this treatment and the stem cell transplant to you in more detail. You will be required to sign a separate consent form.

Study Visits:

One (1) time each month:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests and to check your kidney and liver function.
* You will have an electrocardiogram (EKG -- a test that measures the electrical activity of the heart).

On Day 14 (+/- 2 days) of of Cycle 1, blood (about 2 teaspoons) will be drawn for routine tests and to check your kidney and liver function. You can have this blood drawn at a local lab or clinic that is closer to your home. The results will be sent to the study doctor at MD Anderson.

During Week 2 of Cycle 1, a member of the study staff will call to ask you about any symptoms you may be having. This call should last about 5-10 minutes.

Length of Study:

You will be on study for up to 1 year after the transplant. You may be taken off study early if the disease gets worse, if you have any intolerable side effects, of if you are unable to follow study directions.

Your participation on this study will be over after about 1 year of follow-up tests.

End-of-Study Visit:

Within about 7 days after your last dose of pacritinib, but before your stem cell transplant:

* You will have a physical exam and an ultrasound, MRI, or CT scan of your abdomen to measure your liver and spleen.
* You will have an EKG.

Before your transplant, you will have a bone marrow biopsy/aspiration to check the status of the disease.

Follow-Up Tests:

You will have follow-up visits at about 1, 3, 6, and 12 months after the transplant:

* You will complete 3 questionnaires about your symptoms and quality of life. It should take about 20-30 minutes to complete the questionnaires.
* At Month 3, you will have a physical exam and an ultrasound, MRI, or CT scan of your abdomen to measure your liver and spleen. This will be repeated at Month 12, if your doctor thinks it is needed.
* At Months 3 and 12, you will have a bone marrow biopsy/aspiration to check the status of the disease.

This is an investigational study. Pacritinib is not FDA approved or commercially available. It is currently being used for research purposes only. The study doctor can explain how the study drug is designed to work.

Up to 40 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Idiopathic Myelofibrosis or Myelofibrosis secondary to Polycythemia Vera or Essential Thrombocythemia.
2. Patients 18 years to less than or equal to 70 years.
3. Patients wanting to pursue transplant.
4. Patients must have a Zubrod PS equal or less than 2.
5. Calculated creatinine clearance greater than 50ml/min. using the Cockcroft-Gault equation.
6. Ejection fraction equal or above 40%.
7. Serum direct bilirubin less than 1 mg/dl (unless due to Gilbert's syndrome or hemolysis).
8. SGPT equal or less than 4 x normal values.
9. Corrected DLCO equal or above 50% of expected.
10. Negative Beta HCG test in a woman with childbearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization) and if fertile, males and females must agree to use contraceptives.

Exclusion Criteria:

1. Patients with low risk myelofibrosis.
2. Uncontrolled life-threatening infections.
3. HIV positive.
4. Patients with active viral hepatitis.
5. Prior treatment with Pacritinib.
6. Prior stem cell transplant.
7. QTc greater than 450 ms.
8. CYP3A4 strong or moderate inhibitors/inducers in the past 7 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uday Popat, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Idiopathic Myelofibrosis or Myelofibrosis secondary to Ploycythemia Vera or Essential Thrombocythemia that are 18 to 70 years old that want to pursue a transplant. They start the Pacritinib per-transplant and can proceed to transplant 60 days after starting Pacritinib but no more than 180 days.
Groups:
- Pacritinib Pre- Transplant: Patients will start pacritinib 200 mg po bid and can proceed to transplant after 60 days of starting pacritinib but not more than 180 days
Period: Overall Study
Arm/Group | Pacritinib Pre- Transplant
Started | 4
Completed | 0
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — FDA Clinical hold-patients taken off | 2

BASELINE CHARACTERISTICS:
Groups:
- Pacritinib Pre- Transplant: Patients will start pacritinib 200 mg po bid and can proceed to transplant after 60 days of starting pacritinib but not more than
Arm/Group | Pacritinib Pre- Transplant
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The protocol was to enroll at least 21 evaluable participants, defined as patients who received Pacritinib for >/=60 days but less than 180 days. We enrolled four participants, however all four were not evaluable since no one was able to complete 60 days of Pacritinib.
Time Frame: participants who received Pacritinib for >/= 60 days but less than 180 days who undergo transplant with a matched related or at least 7/8 matched unrelated donor. The protocol was to evaluate progression free survival at one year.
Population: Four participants were not evaluable and no analysis was done.
Arm/Group | Pacritinib Pre- Transplant
Number analyzed (Participants) | 0

2. Other Pre Specified Outcome: Evaluate Safety and Efficacy of Pacritinib.
Description: Evaluate safety and efficacy of this therapy determined by Neutrophil and platelet engraftment, Non-relapse mortality at one year post transplant, Overall survival at one year post transplant, Liver and spleen response to Pacritinib, Immune recovery, quality of life and symptom score, Primary and secondary graft failure,Complete remission, Relapse.
Time Frame: Start of Pacritinib to one year post transplant
Population: Four participants was invaluable and no analysis was done.
Arm/Group | Pacritinib Pre- Transplant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 07/31/2015 to 02/25/2016
Description: The severity of the adverse events (AEs) will be graded according to the Common Terminology Criteria v4.0 (CTCAE). We will not capture expected Grade 1 and Grade 2 AEs. Grade 3 and 4 AEs will be collected and recorded in the medical record. Only Pacritinib-related adverse events and protocol specific data will be entered into PDMS/CORe. PDMS/CORE will be used as the electronic case report form for this protocol.
Arm/Group | Pacritinib Pre- Transplant
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pacritinib Pre- Transplant (N=4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT02410551/Prot_SAP_000.pdf